CLINICAL TRIAL: NCT07381387
Title: Effect of Supra-abdominal Versus Infra-abdominal Muscles Training Combined With LASER on Sternal Instability After Open Heart Surgery
Brief Title: Comparison of Supra-abdominal ex Versus Infra-abdominal With Laser on Median Sternotomy
Acronym: LLL/CABG
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Beni-Suef University (Other)
Responsible Party: Principal Investigator, Mayar Mohammed Khalifa Ahmed, Physiotherapist, Beni-Suef University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: FPTBSUREC/0102/131024; NO secondary ID (Other: NO secondary ID)
Record Dates: First submitted 2025-11-27; First posted 2026-02-02 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Sternal Instability After Median Sternotomy
Keywords: sternal instability

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Group A: Supra-abdominal + LLL (Experimental): Participants in this group receive a combined intervention in addition to the standard cardiac rehabilitation program during phase I
  Interventions: Behavioral: supra abdomen resisted exercises combined with LLL + Traditional cardiac rehabilitation program of phase one; Other: patients will receive Traditional cardiac rehabilitation program of phase one only
- Group B: Infra-abdominal + LLL (Experimental): Participants in this group receive a combined intervention in addition to the standard cardiac rehabilitation program during phase I.
  Interventions: Behavioral: ): patients will infra abdomen resisted exercises combined with LLL +Traditional cardiac rehabilitation program of phase one.; Other: patients will receive Traditional cardiac rehabilitation program of phase one only
- Group C: LLL Only (Experimental): Participants in this group receive low-level laser therapy in addition to the standard cardiac rehabilitation program during phase I.
  Interventions: Other: patients will receive Traditional cardiac rehabilitation program of phase one only
- Group D: Control (Experimental): Participants in this group receive the standard cardiac rehabilitation program during phase I.
  Interventions: Behavioral: patients will receive Traditional cardiac rehabilitation program of phase one with LLL; Other: patients will receive Traditional cardiac rehabilitation program of phase one only

INTERVENTIONS:
Behavioral: supra abdomen resisted exercises combined with LLL + Traditional cardiac rehabilitation program of phase one — Ex 1:- Sitting In Erect Position + Breathing For 3 Min And Repeat 2 Times {Neutral Spine } Ex 2:- Hands On Lower Costal + Inhale Maximally For 5 Sec, Exhale Slowly With Abdominal Muscle Contract And Repeat 10 Times {Thoracic Expansion } Ex 3 :- Hands On Iliac Crest Deep Inhalation + Slow Exhalation For 5 Sec + Contraction Of Abdominal Muscle With Hands Closing At The Hip {Abdominal } Ex 4 :- Inhale Rotate The Trunk To Opposite Side Of Resistance Given By PT + Exhale + Contract Abdominal Muscle { Abdominal Ex With Trunk Rotation } Ex 5:- Cross Arm On Upper Thorax Inhale Raising + Exhale + Contract + While Expiration, Incline Trunk To Opposite Of Resistance Repeat 5 Times For Each Arm Separately Ex6:- Inhale + Raising Two Arm To Shoulder Level With Extended Elbow + Exhale + Contract 5 Sec {Arm - Trunk Dissociation } Repeat 10 Times Ex 7:- Inhale + Flex Arm With Extension Elbow + Exhale + Contract And Return Arm {Alternate Trunk And Shoulder Dissociatio
  Arms: Group A: Supra-abdominal + LLL
Behavioral: ): patients will infra abdomen resisted exercises combined with LLL +Traditional cardiac rehabilitation program of phase one. — Ex 1:- Sitting In Erect Position + Breathing For 3 MinAnd Repeat 2 Times Ex 2:- Hands On Lower Costal + Inhale Maximally For 5 Sec, Exhale Slowly With Abdominal Muscle Contract And Repeat 10 Times Ex 3 :- Hands On Iliac Crest Deep Inhalation + Slow Exhalation For 5 Sec + Contraction Of Abdominal Muscle With Hands Closing At The Hip Ex 4 :- Inhale Rotate The Trunk To Opposite Side Of Resistance Given By PT + Exhale + Contract Abdominal Muscle Ex 5:- Cross Arm On Upper Thorax Inhale Raising + Exhale + Contract + While Expiration, Incline Trunk To Opposite Of Resistance Repeat 5 Times For Each Arm Separately Ex 6 :- Inhale + Raise Knee With Flexed Hip + Expiration + Contract Ex 7: Inhale + Exhale + Adducting Hip And Knees + Contract Ex 8 :- Inhale + Raise One Knee + Exhale+Contract+Trunk Rotation To The Side Of Raised Leg
  Arms: Group B: Infra-abdominal + LLL
Behavioral: patients will receive Traditional cardiac rehabilitation program of phase one with LLL — A probe laser device will be usedat median sternotomy site. at a distance of 2 cm from each other, for a total of five to eight points. the device will be placed in a perpendicular position to the sternum each spot for 60 sec for a total session time of 5-10 min. Each patient will receive one session daily, three times a week, for four consecutive weeks:•Treatment time per point (s) 60•Laser beam Class :3B•Laser Type :Semiconductor GaA.Modes of Operation :Continuous Pulse upto 5 khz.•Wave Length: 685nm•Maximum Probe Power: 500 mw•Power Density:0.8w/cm2•Max Energy within 1 min 2.4 Joules•Number of spots 8 Patients will be instructed to perform deep breathing using incentive spirometry in the form of four sets, each consisting of 10 deep breaths for a total of 40 deep breaths, with a hold at the end of inspiration, then huffs and coughs with the support of pillows at the incision. The patients will be instructed to follow sternal precautions
  Arms: Group D: Control
Other: patients will receive Traditional cardiac rehabilitation program of phase one only — Patients will be instructed to perform deep breathing using incentive spirometry in the form of four sets, each consisting of 10 deep breaths for a total of 40 deep breaths, with a hold at the end of inspiration, then huffs and coughs with the support of pillows at the incision. The patients will be instructed to follow sternal precautions

SUMMARY:
the aim of this study is to find out the differences between the effect of supra- abdomen exercises and the effect of infra-abdomen exercise combined with LASER And the effect of LOW LEVEL LASER only on sternal instability. Methods: 120 patients of both sexes who had acute sternal instability post-open heart surgery will be recruited in this study at Assiout University Hospitals; their ages will be > 18 years. They will be randomly assigned into 4 equal groups:

1. Study group (A): patients will receive supra-abdominal resisted exercises combined with LLL and the traditional cardiac rehabilitation program of phase one.
2. Study group (B): patients will do infra-abdominal resisted exercises combined with LLL and the traditional cardiac rehabilitation program of phase one.
3. Study group (c): patients will receive a traditional cardiac rehabilitation pro-gram of phase one with LLL
4. Control group: patients will receive the traditional cardiac rehabilitation pro-gram of phase one only

DETAILED DESCRIPTION:
Type of study: Randomized controlled trial This study is a prospective interventional study one that will be conducted on 120 patients of both sexes who had acute sternal instability post-open heart surgery; their ages will be < 18 years. They will be recruited from Assiut University Hospitals and will randomly be divided into 4 equal groups

1. Study group (A): patients will receive supra-abdomen resisted exercises combined with LLL and the traditional cardiac rehabilitation program of phase one.
2. Study group (B): patients will do infra-abdomen resisted exercises combined with LLL and the traditional cardiac rehabilitation program of phase one.
3. Study group (c): patients will receive a traditional cardiac rehabilitation pro-gram of phase one with LLL
4. Control group: patients will receive Traditional cardiac rehabilitation pro-gram of phase one only

ELIGIBILITY:
IInclusion criteria :

All included patients will be:

* Their age 18<.
* Both sexes.
* Hemodynamic stable.
* Acute sternal instability.
* Able to provide informed consent.

Exclusion criteria:

Patient will be excluded if:

* Emergency or urgent operation.
* Revision sternotomy.
* Manifesting hypoxemia.
* Partial oxygen pressure in arterial blood < 60 mmHg.
* Renal insufficiency with serum creatinine ≥ 1. 8 mg/dl after surgery.
* Low cardiac output syndrome with ST segment elevation in multiple electrocardiogram leads.
* Cardiac arrhythmias or hypotension.
* Other medical conditions, such as diabetes, uncontrolled hypertension and obesity.
* Previous medical history including conditions that may have influenced the provision of physiotherapy interventions, such as severe asthma, chronic airflow limitation, bronchiectasis, ankylosing spondylitis or lumbar disc prolapse.
* Impaired cognition.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2026-01-27 (Estimated); Primary Completion 2026-07-27 (Estimated); Study Completion 2026-07-27 (Estimated)

PRIMARY OUTCOMES:
sternal instability | at baseline and after finishing program (up to one month)
  1. Sternal separation measurement: The ultrasound unit head was adapted by fixing it to a microphone stand to facilitate contact with the chest of a seated subject. The amount of sternal separation at different vertical points on the sternum could now be measured from the projected image using the proprietary software for the unit
  2. Sternal instability scale:
     * Grade 0:
     * Clinically stable sternum, no detectable motion (normal).
     * Grade 1:
     * Minimally separated sternum with a slight increase in motion upon special testing (upper limbs, trunk).
     * Grade 2:
     * Partially separated sternum, regional with moderate increase in motion upon special testing.
     * Grade 3:
     * Completely separated sternum along the entire length with marked increase in motion upon special testing.

SECONDARY OUTCOMES:
Functional Impairment Scale: | at baseline and after finishing program (up to one month)
  1)Functional Impairment Scale: Functional impairment was based on a numerical scale from 0 to 10, as follows: 0-3, did not interfere with activities; 4-6, interfered but did not prevent activities; 7-9, prevented activities; and 10, prevented activities and/or caused lack of control Higher scores indicate greater functional impairment.
pain assessment | at baseline and after finishing program (up to one month)
  Pain intensity will be measured using the Visual Analog Scale (VAS), a 10-cm horizontal line ranging from 0 to 10, where 0 represents no pain and 10 represents the worst imaginable pain. Participants will be asked to mark the point that best reflects their perceived pain intensity. Higher scores indicate greater pain intensity.
The Activity Status Index for Duke | at baseline and after finishing program (up to one month)
  Functional capacity will be assessed using the Duke Activity Status Index (DASI), a self-reported 12-item questionnaire that evaluates the ability to perform daily physical activities and estimates functional capacity in metabolic equivalents (METs). Scores range from 0 to 58.2, with higher scores indicating better functional capacity.

CONTACTS AND LOCATIONS:
Overall Officials: SHERIN HASSAN MOHAMMED MEHANI. MEHANI., professor, Principal Investigator — benisueif university; MOHAMMED AHMED KHALIL SALAMA SALAMA, professor, Principal Investigator — Assiut University
Locations (1):
- مستشفي القلب الحامعي -مستشفيات جامعه اسيوط, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: No